CLINICAL TRIAL: NCT02906891
Title: A Pilot Study of Nocturnal Hypoglycemia Prevention in Type 1 Diabetes Using the Vigilant Diabetes Management Companion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources to complete study
Sponsor: InSpark Technologies, Inc. (Industry)
Collaborators: East Carolina University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VG2NOCHPUS1
Record Dates: First submitted 2016-02-19; First posted 2016-09-20 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Hypoglycemia; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Usual Care Patients on MDI or CSII (Experimental): Usual Care Patients on MDI or CSII Usual care patients on multiple daily injections of insulin (MDI) or insulin pumps (CSII) will be their own controls against baseline and will use the Vigilant Diabetes Management Application in conjunction with a wireless blood glucose meter for three months.
  Interventions: Device: Vigilant Diabetes Management Application

INTERVENTIONS:
Device: Vigilant Diabetes Management Application — The Vigilant Diabetes Management Companion by InSpark Technologies was developed to assist in the prevention of hypoglycemia by providing the individual with an unobtrusive analysis of their blood glucose values and notifying them about periods of upcoming risk for low and high blood glucose; and in particular periods of risk for severe hypoglycemia. This allows the individual to take preventive corrective action. Subjects will download the Vigilant DiabetesManagement Application and use it in conjunction with a study supplied wireless blood glucose meter. They will check blood glucose values at least three times a day and receive summaries and notifications from Vigilant regarding periods of risk and blood glucose patterns.
  Other Names: Vigilant

SUMMARY:
A single center pilot study assessing the Vigilant Diabetes Management Companion for the prevention of recurrent nocturnal hypoglycemia in type I diabetes patients.

DETAILED DESCRIPTION:
This is a pilot study to determine whether a large-scale randomized trial is feasible. The pilot study will test if the Vigilant Diabetes Management System is effective in adults with T-I Diabetes in preventing nocturnal hypoglycemia, improving moderate hypoglycemia, improving diabetes quality of life and in reducing fear of hypoglycemia.

2ndary aim: Health care professional adoption of the technology - medication titrated or changed, reports that the system facilitated treatment decisions, provided meaningful feedback and or reduced time.

This is a single center 12-week Pilot trial with one arm. Subjects will serve as their own controls. The study will include usual care patients on MDI (multiple daily injections) or CSII (continuous subcutaneous insulin infusion) with the additional use of the Vigilant Diabetes Management System. There will be a 4-week baseline period prior to the 12-week intervention. Subject participation for the 4-week baseline period will last for 2 to 4 hours during two visits. Subjects participating in the intervention phase of 12 weeks will require one additional visit for 2 to 3 hours at 3 months, which is routine for this population.

Participants will be provided with a wireless blood glucose meter for the duration of the study and will download the Vigilant mobile application to their mobile phone.

The Vigilant system stores blood glucose test results, pattern events, and user settings. In addition to receiving blood glucose measurements entered from the user, storing and displaying them, Vigilant provides the following features and tools for the user:

Blood Glucose Reading review and editing: The user will be able to review data logs and manually edit blood glucose results.

Pattern Messages: Alerts the user that one or more patterns were found in the results that were entered, including patterns that are indicative of risk of severe hypoglycemia in the next 24 hours.

Long Term Control Summary: Identifies the current and retrospective blood glucose averages and variability.

The following blood glucose patterns will be identified by the Vigilant application:

Weekly and monthly glucose averages overall and within daily time periods Daily periods of infrequent testing Daily periods of high, low or variable blood glucose - Daily Pattern Messaging System.

Patterns of blood glucose indicative of increased risk of low blood glucose levels in the next 24 hours - Hypo Risk Indicator.

Weekly and monthly blood glucose variability - Average Daily Risk Range or ADRR.

Vigilant incorporates a Tutorial Mode which offers detailed feedback on the meaning of pattern analyses performed by the software. In addition, two separate training videos have been developed for patients and clinicians to initiate them on use and understanding of the device and its features.

Caregivers will have access to the information outlined above, as well as summary screens that highlight glycemic control metrics and patients and risk notifications for all of their patients on Vigilant, subject to patient approval.

Subjects will be recruited from one diabetes clinic. Patients with type I diabetes and a history of nocturnal and or severe hypoglycemia will be assessed to see if they are eligible for the study. All those who are considered eligible will be approached to give their written, informed consent before attending a screening visit where the inclusion criteria will be checked.

At the Screening Visit the following procedures will be performed and criteria will be checked and documented:

Signed and dated informed consent Assignment of subject number Inclusion and exclusion criteria Demographics - date of birth, gender, race and ethnicity Subjects Diabetes history Clinician Professional history SMBG-self-monitoring of blood glucose training with study meter Use of study hypoglycemia diary Completion of study questionnaires

After consent, participants will participate in the 4-week run-in baseline period before the 12-week pilot intervention to collect baseline data on glycemic control and hypoglycemia and to assess adherence with testing criteria. All participants will be asked to conduct SMBG or self-monitoring of blood glucose three or more times a day and asked to record the clinical details of any hypoglycemia events.

At the end of the 4-week baseline period, participants will return for a study visit where the investigator will complete the following:

Download the SMBG and hypoglycemia diary and data Obtain A1C Affirmation of participant commitment to test and record To continue in the study, subjects will need to have obtained at least three blood glucose values per day and have recorded hypoglycemia symptoms and episodes.

Prior to the 12-week intervention period, all study participants will complete validated study questionnaires -Hypoglycemia Fear, Diabetes Empowerment Survey etc.

At visit 2, the subjects will complete training with the Vigilant program. They will watch a video demonstration on an iPhone , Android or iPod Touch that explains the use of the Vigilant device. Study participants will be provided a wireless blood glucose monitor and asked to follow their normal diabetes management program for the subsequent 12 weeks.

They will be asked to use the Vigilant program at home in conjunction with the provided wireless meter for the subsequent 12 weeks, according to the following instructions:

The subject will follow their typical blood glucose-testing regimen, with the exception that they must perform an average of at least 3 fingerstick blood glucose measurements daily during that time.

Subjects will be asked to keep a log of HRI or hypoglycemia risk indicator pattern messages received, with any entered glucose reading if delivered at that time, and what diabetes management action they chose to perform when the message is received.

Subjects will be asked to log whether or not they understand the feedback given, and what action is taken to address the pattern, if any.

Subjects will not be required to perform any specific diabetes management action to address identified patterns. Worksheets will be provided to patients to facilitate record keeping for pattern message feedback.

It is preferred that the subject use predominantly the study supplied meter during the course of the 12 weeks of home use and only two glucometers maximum.

Subjects will be instructed to change the date and time of their meter in the event of any changes for daylight savings time, or travel to different time zones, so that it matches the iPod touch or Phone clock time.

Subject will be instructed on proper SMBG technique including using water and dry towel prior to testing, avoiding alternate site testing, and using the second hanging blood drop. The subject will be asked to demonstrate an SMBG test at the visit to document proper technique.

Participants will be followed up at three months during the 12-week intervention period. Subjects will also receive a telephone or email communication from the study manager within several days of the beginning of the home use portion of the study to ensure the patient understands the protocol and is entering data according to instructions. At this time they will also be asked to send several screen shots of their application with a log of their data and patterns that have been identified, to ensure the device is working according to the intended use and data is being entered.

Another follow up will occur 4 weeks into the study where the patients will be asked the same questions and given the same instructions.

Subjects involved in this study should also allow their Vigilant-using clinician to see their Vigilant patterns, and also plan to see their Vigilant-using clinician at least once for a regular check up during their Vigilant use period. This can be done at Visit 3, if desired.

A follow-up and final visit will occur at the three-month end of the 12 week intervention period, which is the typical routine schedule for usual care. Additional visits may be scheduled by provider as indicated for diabetes management.

The following procedures will be performed in at the follow-up visit:

Blood draw for HbA1c Download SMBG data Review of patient diaries and data Data collection of hypoglycemia and other events Review of Vigilant pattern messages and patient log Completion of study questionnaires and surveys

ELIGIBILITY:
Inclusion Criteria:

* • Male or female participants aged between 18 and 75 years

  * Clinical diagnosis of type 1 diabetes mellitus and using multiple daily injections or CSII for at least six months
  * Patient has had documented nocturnal hypoglycemia in the last 2 months with an associated blood sugar reading less than 56mg/dL. Night is defined as the 8 hour interval when the patient usually sleeps (I.e. 11:00 pm to 7:00 am, for example).

OR

* Patient has had at least 1 severe low at night in the last 6 months (helped by another). Night is defined as the 8 hour interval when the patient usually sleeps (I.e. 11:00 pm to 7:00 am, for example).
* Willing to monitor and record signs and symptoms of hypoglycemia
* Willing to test blood glucose levels at least three times a day
* Ability to use Android or IOS mobile phone
* No CGM Users

Exclusion Criteria:

* • Pregnancy

  * Unable to use the technology
  * Any condition that in the investigators judgment is likely to cause the participant to be unable e to understand or provide informed consent
  * Unwilling to use SMBG at least three times a day
  * Unwilling to monitor and record signs and symptoms of hypoglycemia
  * Individuals who are unwilling to share their glucose meter data

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Reduction in the aggregate rate of nocturnal biochemical severe hypoglycemia in the Vigilant period versus the Baseline period as measured by meter or logged blood glucose values (mg/dL). | 3 months
  Nocturnal biochemical severe hypoglycemia is defined by 1) a reading below 56 mg/dL at night OR 2) a severe low (requires assistance from another) at night. Night is defined as the 8 hour interval when the patient usually sleeps (ie. 11:00pm to 7:00 am, for example). Baseline is defined as collected glycemic data prior to Vigilant initiation as well as the run-in period.
Reduction in the aggregate rate of nocturnal hypoglycemia in the Vigilant period versus the Baseline period as measured by meter or logged blood glucose values (mg/dL). | 3 months
  Nocturnal hypoglycemia is defined by 1) a reading below 70 mg/dL at night OR 2) a severe low (requires assistance from another) at night.Night is defined as the 8 hour interval when the patient usually sleeps (I.e. 11:00 pm to 7:00 am, for example).
  Night is defined as the 8 hour interval when the patient usually sleeps (ie. 11:00pm to 7:00 am, for example. Baseline is defined as collected glycemic data prior to Vigilant initiation as well as the run-in period.

SECONDARY OUTCOMES:
An aggregate (total study population) reduction in the rate of mild hypoglycemia (biochemical and logged) as measured by home blood glucose values <70 mg/dL at 3 months, compared to the monthly rate of hypoglycemia in the Baseline period. | 3 months
  Logged values will only be considered in the calculation if no duplicate hypoglycemic readings within 15 minutes of the logged value can be found in the patient's meter download data.
An aggregate reduction in the rate of biochemical severe hypoglycemia as measured by home blood glucose values <40 mg/dL, during months 1-3, compared to the monthly rate of biochemical severe hypoglycemia in the Baseline period. | 3 months
  biochemical and logged) Logged values will only be considered in the calculation if no duplicate hypoglycemic readings within15 minutes of the logged value can be found in the patient's meter download data.
An aggregate reduction in average HbA1will be measured at baseline using DCA 2000 or equivalent NGSP- certified point-of-care method or local laboratory at 3 months, compared to HbA1c levels obtained at study initiation. | 3 months
  Reduction in HbA1c in three months vs baseline period.
An aggregate reduction in the survey self-reported rate of use of; 1) Glucagon 2) Emergency medical services for hypoglycemia, and 3) Hospital, urgent care or clinic visits for hypoglycemia or associated with hypoglycemia care visits. | 3 months
  Reduction in Glucagon use, Emergency services use, Hospitalizations and or ER/Urgent Care visits for hypoglycemia events vs baseline. In the intervention period, compared to the rate in the 3 month period prior to study initiation. Total study population data will be obtained from adding up the number of incidents on the self-reported surveys. In the event that additional data on emergency medical services, hospital, urgent care or clinical visits is available through the clinician of the patient, or through the patient's health plan or insurance, and the patient elects to provide this information for the benefit of the study, these records will be used to verify and / or supplement occurrences. Any record discrepancy will be resolved at the discretion of the principal investigator
An aggregate reduction in the mean glycemic variability, as measured by monthly ADRR (Average Daily Risk Range), calculated based on downloaded meter download data | 3 months
  Reduction in glycemic variability using the ADRR measure vs baseline period at 3 months, compared mean monthly ADRR value based on meter downloads at the end of the baseline period.
An aggregate (total study population) reduction in the LBGI and HBGI, as measured by percent of readings in and out of range calculated based on downloaded blood glucose meter download data. | 3 months
  Reduction in LBGI and HBGI in the three month intervention period versus baseline. In range = 70-180 mg/dL, Out of range is < 70 and > 180 mg/dL). At 3 months, compared to mean monthly percent of readings in and out of range based on blood glucose meter downloads at the end of the baseline period.
Reduction in reported fear of hypoglycemia as compared to baseline Fear of Hypoglycemia Fear Survey. The Hypoglycemia Fear Survey II (HSF II) will be used. | 3 months
  Reduction in reported fear of hypoglycemia and improvement in quality of life as compared to baseline survey results. It is a validated scale that consists of questions that measure behaviors involved in avoidance and over treatment of hypoglycemia and a worry subscale that measures anxiety and fear surrounding hypoglycemia. The Hypoglycemic Fear Survey endpoint will be met if the average ratings across all survey questions will be improved at 3 months, versus at study initiation.
  Exploratory analyses of the association of Hypoglycemia Fear Survey answers and clinical improvement will be done at the discretion of the Principal Investigator and Sponsor
Improvement in self-reported lost work productivity as a result of hypoglycemia. Individuals will complete a questionnaire about lost work days as a result of hypoglycemia at baseline and at 3 months. | 3 months
  Improvement in lost work productivity as a result of hypoglycemia as compared to self reported baseline survey results.
Improvement in self-reported psychosocial self-efficacy as compared to baseline measured using the Diabetes Empowerment Scale Short Form (DES-SF). | 3 months
  Improvement in self reported diabetes psychosocial self-efficacy. The Diabetes is an abbreviated, validated scale of the Diabetes Empowerment Scale (DES), which was developed and validated by the Michigan Diabetes Research Center for the measurement of psychosocial self-efficacy of people with diabetes.

OTHER OUTCOMES:
Average ratings of "acceptable" or better from self-reported survey clinician feedback on the utility of Vigilant in managing patients. | 3 months
  The secondary endpoint for clinicians will be met with average ratings of "acceptable" or better from self- reported clinician feedback on a survey on the utility of Vigilant in managing patients in their practice; supporting medication titration, facilitating positive treatment decisions, providing meaningful feedback and reducing time spent doing data analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Fuqua, RN, MSN, Study Chair — InSpark Technologies, Inc.; Robert Tanenberg, MD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] ter Braak EW, Appelman AM, van de Laak M, Stolk RP, van Haeften TW, Erkelens DW. Clinical characteristics of type 1 diabetic patients with and without severe hypoglycemia. Diabetes Care. 2000 Oct;23(10):1467-71. doi: 10.2337/diacare.23.10.1467. PMID 11023138
- [Result] Epidemiology of severe hypoglycemia in the diabetes control and complications trial. The DCCT Research Group. Am J Med. 1991 Apr;90(4):450-9. PMID 2012085
- [Result] Cryer PE, Gerich JE. Glucose counterregulation, hypoglycemia, and intensive insulin therapy in diabetes mellitus. N Engl J Med. 1985 Jul 25;313(4):232-41. doi: 10.1056/NEJM198507253130405. PMID 2861565
- [Result] Ha WC, Oh SJ, Kim JH, Lee JM, Chang SA, Sohn TS, Son HS. Severe hypoglycemia is a serious complication and becoming an economic burden in diabetes. Diabetes Metab J. 2012 Aug;36(4):280-4. doi: 10.4093/dmj.2012.36.4.280. Epub 2012 Aug 20. PMID 22950059
- [Result] Otto EA, Tannan V. Evaluation of the utility of a glycemic pattern identification system. J Diabetes Sci Technol. 2014 Jul;8(4):830-8. doi: 10.1177/1932296814532210. Epub 2014 May 12. PMID 24876425
- [Result] Kovatchev BP, Otto E, Cox D, Gonder-Frederick L, Clarke W. Evaluation of a new measure of blood glucose variability in diabetes. Diabetes Care. 2006 Nov;29(11):2433-8. doi: 10.2337/dc06-1085. PMID 17065680
- [Result] Kovatchev BP, Mendosa P, Anderson S, Hawley JS, Ritterband LM, Gonder-Frederick L. Effect of automated bio-behavioral feedback on the control of type 1 diabetes. Diabetes Care. 2011 Feb;34(2):302-7. doi: 10.2337/dc10-1366. Epub 2011 Jan 7. PMID 21216860
- [Result] Edelman SV, Blose JS. The Impact of Nocturnal Hypoglycemia on Clinical and Cost-Related Issues in Patients With Type 1 and Type 2 Diabetes. Diabetes Educ. 2014 May;40(3):269-279. doi: 10.1177/0145721714529608. Epub 2014 Apr 2. PMID 24695260